CLINICAL TRIAL: NCT01284530
Title: Evaluation of the Pharmacokinetics, Safety, and Tolerability of TPM XR as Adjunctive Therapy in Pediatric Subjects With Epilepsy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Supernus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 538P107
Record Dates: First submitted 2011-01-25; First posted 2011-01-27 (Estimated); Last update posted 2016-06-02 (Estimated); Status verified 2016-05

CONDITIONS: Epilepsy
Keywords: Epilepsy; Pediatrics; Young Adults
MeSH Terms: conditions — Epilepsy

ARMS (4):
- Conversion-25 (Experimental): 25 mg
  Interventions: Drug: TPM XR
- Conversion-50 (Experimental): 50 mg
  Interventions: Drug: TPM XR
- Conversion-100 (Experimental): 100 mg
  Interventions: Drug: TPM XR
- Conversion-200 (Experimental): 200 mg
  Interventions: Drug: TPM XR

INTERVENTIONS:
Drug: TPM XR — Equivalent TDD in XR form, QD, Day 1-14

SUMMARY:
Multidose, Open-label, Multi-center Study to examine the steady state pharmacokinetics of TPM XR, as well as, safety and tolerability of repeated oral dosing in pediatric subjects with epilepsy.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide written IAF, as appropriate, with written informed permission (including ICF where required by regional laws or regulations) from the parent or LAR.
2. Male or female aged 4 to 17 years, inclusive, with a current diagnosis of partial onset or primary generalized epilepsy.
3. Current AED therapy including a stable dose of TPM IR as either adjunctive or monotherapy. All AED therapy (including a Vagal Nerve Stimulator) must have been initiated more than one month prior to Visit 1 and doses must be stable for at least two weeks prior to Visit 1.
4. No diagnosis of a progressive neurological disorder based on previous imaging.
5. Weight within the 25 - 80% weight-for-age percentiles based on the National Center for Health Statistics Growth Charts, and not less than 15.0kg.
6. Able and willing to swallow whole capsules.
7. FOCP should either be sexually inactive for two weeks prior to the first dose and throughout the study or, if sexually active, will be using an effective birth control method.

Exclusion Criteria:

1. A documented history of status epilepticus in the past year or seizures secondary to conditions other than epilepsy.
2. Use of either phenytoin or carbamazepine as current AEDs.
3. Diagnosis or an electroencephalogram consistent with a diagnosis of seizure disorders other than partial onset or primary generalized epilepsy.
4. Current diagnosis of Major Depressive Disorder or any history of suicide intent and/or attempt.
5. History or presence of clinically significant, chronic medical condition which, in the opinion of the Investigator, would preclude the subject from entering the study.
6. History of substance abuse or dependence.
7. Females who are pregnant or lactating.
8. Use of an investigational drug or device or participation in an investigational study within 30 days prior to the first dose of SM.

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2011-01; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
steady-state pharmacokinetics (PK) of TPM XR and to assess the safety and tolerability | 14 days
  Relating to repeated oral dosing

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Stocks, Study Director — Supernus Pharmaceuticals
Locations (10):
- United States (10):
  - Sacramento, California
  - Loxahatchee Groves, Florida
  - Miami, Florida
  - Wichita, Kansas
  - Louisville, Kentucky
  - Hackensack, New Jersey
  - Akron, Ohio
  - Dallas, Texas
  - Norfolk, Virginia
  - Richmond, Virginia